CLINICAL TRIAL: NCT02837523
Title: Biomarker for Cystinosis Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Cystinosis Disease: BioCystinosis (BioCystinosis)
Acronym: BioCystinosis
Status: Withdrawn | Type: Observational
Why Stopped: No longer pursued
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BCY 06-2018
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Renal Fanconi Syndrome; Photophobia; Hypophosphatemia
Keywords: Cystinosis Disease; Biomarker
MeSH Terms: conditions — Fanconi Syndrome; Photophobia; Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, maximal 7,5 ml of blood will be taken via using a dry blood spot filter card. To proof the correct Cystinosis diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Cystinosis disease will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with a Cystinosis disease or high-grade suspicion for Cystinosis disease

SUMMARY:
Development of a new mass spectrometry-based biomarker for the early and sensitive diagnosis of Cystinosis disease from the blood

DETAILED DESCRIPTION:
Cystinosis is a rare, multisystem genetic disorder characterized by the accumulation of an amino acid called cystine in different tissues and organs of the body including the kidneys, eyes, muscles, liver, pancreas and brain. Generally, Cystinosis is broken down into three different forms known as nephropathic Cystinosis, intermediate Cystinosis and non-nephropathic (or ocular) Cystinosis. Early detection and prompt treatment are critical in slowing the development and progression of symptoms associated with Cystinosis. The kidneys and eyes are the two organs most often affected. Individuals with nephropathic or intermediate Cystinosis ultimately require a kidney transplant. Non-nephropathic Cystinosis only affects the corneas of the eyes. Cystinosis is caused by mutations of the CTNS gene and is inherited as an autosomal recessive disease.

The specific symptoms and severity of Cystinosis vary greatly from one person to another based upon several factors including age of onset and whether the disorder is promptly diagnosed and treated. The progression of the disorder can be slowed by early diagnosis and treatment. Eventually, Cystinosis can affect all tissues of the body. The age of onset for different symptoms varies greatly.

• NEPHROPATHIC CYSTINOSIS (renal Fanconi disease)

Nephropathic Cystinosis is the most frequent and most severe form of Cystinosis. The symptoms of nephropathic Cystinosis usually become apparent within the second half of the first year of life.

Growth failure and renal Fanconi disease are usually the first noticeable complications of the disorder. Although infants appear normal at birth, by the age of one they often fall into the third percentile for height and weight. In addition, affected infants may have episodes of vomiting, poor appetite, and feeding difficulties that contribute (along with kidney dysfunction) to nutritional deficiency and the failure to gain weight and grow at the expected rate (failure to thrive). Ultimately, growth in untreated children with Cystinosis occurs at 60 percent the expected rate.

Infants with nephropathic Cystinosis develop renal Fanconi disease, a rare disorder characterized by kidney dysfunction. The kidney tubules fail to reabsorb a variety of needed substances, including the compounds mentioned above as well as amino acids, phosphate, calcium, glucose, carnitine, certain proteins and electrolytes.

Symptoms of renal Fanconi disease usually become apparent between 6 and 12 months of age and may include excessive thirst (polydipsia), excessive production and passage of urine (polyuria), electrolyte imbalances, vomiting, and dehydration.

Children with nephropathic Cystinosis may also develop symptoms unrelated to the kidneys (extrarenal symptoms). Again, these findings are highly variable and affected children will not develop all of the symptoms discussed below. Specific extrarenal symptoms will vary greatly depending upon the age that treatment is begun and the specific organs that become involved; those organs can include the eyes, bone marrow, liver, pancreas, spleen, intestine, brain, thyroid, muscles and testes.

Affected children may also develop deficiency of thyroid hormone production (hypothyroidism) due to cystine crystals accumulating in the thyroid. Symptoms of hypothyroidism are highly variable, but may include fatigue, feeling cold, dry skin, constipation and depression. Children with nephropathic Cystinosis do not produce tears, sweat or salivate normally. Tear production may be diminished causing the eyes to dry out.

The increased longevity of individuals with nephropathic Cystinosis has revealed that additional complications affecting organs other than the kidneys can occur later during life. These complications develop due to the chronic accumulation of cystine crystals in individuals who have not been adequately treated by cysteamine, although they have undergone a kidney transplant. These additional complications generally develop between 20 and 40 years of age. Accumulation of cystine in muscle tissue can cause muscle dis- ease (myopathy) leading to progressive weakness and wasting of affected muscles. Impairment of muscles in the throat can lead to swallowing and feeding difficulties. Involvement of chest muscles can result in pulmonary insufficiency.

A wide variety of gastrointestinal symptoms can develop including enlargement of the liver (hepatomegaly) causing high blood pressure of the main vein of the liver (portal hypertension), enlargement of the spleen (splenomegaly), gastroesophageal reflux, ulcers, inflammation of the esophagus (esophagitis), and dysfunction of the muscles of the gastrointestinal tract (dysmotility). Additional symptoms include inflammatory bowel disease, tearing of the bowel causing the contents of the intestines to flow into the abdominal cavity (bowel perforation), and inflammation of the peritoneum (peritonitis), which is the membrane that lines the abdominal wall and organs.

Additional findings include metabolic bone disease and an inability to properly digest food due to a lack of digestive enzymes normally produced by the pancreas (pancreatic exocrine insufficiency).

At any age, children may develop an abnormal sensitivity to light (photophobia) and irritation due to the formation of cystine crystals in the cornea. Adults with Cystinosis may also develop abnormalities affecting the eyes including spasms of the eyelids (blepharospasm), band keratopathy and pigmentary retinopathy. Band keratopathy refers to the accumulation of calcium deposits in a band across the central surface of the cornea, which can cause pain and decreased clarity of vision (visual acuity). Pigmentary retinopathy is characterized by progressive degeneration of the retina, the thin layer of nerve cells that line the inner surface of the back of the eyes. Pigmentary retinopathy can impair night and color vision and, eventually, can contribute to overall reduced clarity of vision.

Individuals with nephropathic Cystinosis appear to have a higher rate of diabetes than the general population because of destruction of the pancreas by cystine accumulation.

• INTERMEDIATE CYSTINOSIS

Also known as nephropathic juvenile Cystinosis or adolescent Cystinosis, this form of Cystinosis is characterized by all of the signs and symptoms of nephropathic Cystinosis described above. However, onset of these symptoms does not occur until later perhaps around 8 years of age. Generally, the symptoms are less severe than in the classical infantile nephropathic form and have a slower progression. If untreated, end-stage renal failure in intermediate Cystinosis usually develops at some point between 15 and 25 years of age. There is a spectrum of disease severity in Cystinosis, with overlap of the in-fantile and intermediate forms.

• NON-NEPHROPATHIC CYSTINOSIS

Also known as ocular or "benign" Cystinosis, this form usually affects adult's during middle age; it was once called adult Cystinosis. Kidney disease does not occur in these individuals. The disorder appears to only affect the eyes. Untreated individuals with non- nephropathic Cystinosis eventually develop photophobia due to cystine crystal accumulation in the eyes.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study re- lated procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of the Cystinosis disease or a high-grade suspicion for the Cystinosis disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

Positive family anamnesis for Cystinosis disease

Renal Fanconi syndrome

Photophobia

Hypophosphatemia

Decreased hair and skin pigmentation

Cystine crystals in the cornea

EXCLUSION CRITERIA

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both genders younger than 2 months
* No diagnosis of Cystinosis disease or no valid criteria for profound suspicion of a Cystinosis disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a Cystinosis disease or high-grade suspicion for Cystinosis disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Cystinosis disease from the blood | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  The goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided